CLINICAL TRIAL: NCT03024333
Title: Effect of Different Viscous Foods and Liquids on Swallowing Sounds
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0782-16-EP
Record Dates: First submitted 2017-01-07; First posted 2017-01-18 (Estimated); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Deglutition Disorder
Keywords: Dysphagia; Swallowing Sound; Acoustic Analysis
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy subjects: Healthy subjects are:
  1. Between 19-60 years old
  2. Able to sign the informed consent after the whole study is explained to them
  3. Self-reporting no history of swallowing disorders, neurological deficits and/or cancer of the mouth, neck or brain, or head or neck surgery
  4. Able to sit upright with or without back support of chair
  5. No other diseases affect swallowing function

INTERVENTIONS:
Other:  — Investigators will use the blender to prepare different viscous foods and liquids. Then, a sound detection device will be attached on the participant's neck. The device will record three times of swallowing sounds at three placements (Apleft, Apright, B) separately with participants' head-trunk in neutral position and also record sounds in the neck such as breathing sound, throat clearing and cough sounds. Participants will use 5 ml spoon to intake different viscous foods or liquids. The conversation will also be recorded using a Sony recorder (ICD-SX713) in each data collection session. The voice recording will not be analyzed, which only provides the additional information about which foods or liquids subjects swallow or at which placement sensor records swallowing sounds.
  Other Names: Sony recorder (ICD-SX713); XJ-14402C, Mainstays,Walmart Inc.,Bentonville,AR72716

SUMMARY:
This study is aimed to establish and identify the normal pattern of swallowing sounds and analyze swallowing sounds of different textured foods and viscous liquids in healthy subjects to provide clinical evidence to update dysphagia patients' food.

DETAILED DESCRIPTION:
Upon accepted and consented, the investigators will measure the neck circumference, height and weight of all participants. Then, a sound detection device (iASUS NT3-R Throat Mic Headset, CA, USA) will be attached on the participant's neck. This non-invasive and lightweight (2.3oz) device will record sound vibration signals using a pair of 20mm-diameter sound sensors. The device will record three times of swallowing sounds at three placements (Apleft, Apright, B) separately with participants' head-trunk in neutral position and also record sounds in the neck such as breathing sound, throat clearing and cough sounds. (Apleft, Apright) is the intersection of lateral border of trapezius muscle and intermediate line between the third and fourth cervical vertebrae in the posterior neck region. B is at the lateral cricoid cartilage in the anterolateral neck. Participants will use 5ml spoon to intake foods or liquids at room temperature.

Healthy subjects will conduct the research in the Student Living Center Room 1036/1041 at UNMC. Healthy subjects will be required to swallow different consistency liquids and foods with their head-trunk in neutral position. Participants will also perform one of the following randomly after swallowing foods or liquids: throat clearing after coughing or cough after throat clearing. Before subjects start swallowing test, subjects can try several times if subjects want.There will be 2 sections to complete the whole process. Each section will take 2 hours.The device will record three times of swallowing sounds of each foods and liquids at three placements (Apleft, Apright, B) separately with participants' head-trunk in neutral position.The foods and liquids preparation are also listed at the end of this section.The PI and faculty advisor of the research team will be present during recording swallowing session.

The sound detection device will record sounds which occur in the neck such as swallowing sounds, breathing sound, talking sounds, throat clearing and cough sounds when dysphagia patients intake foods and drinks. The conversation will also be recorded using a Sony recorder (ICD-SX713) in each data collection session.The voice recording will not be analyzed, which only provides the additional information about which foods or liquids subjects swallow or at which placement sensor records swallowing sounds. Recordings will be saved as digital sound wave files and segmented into individual anonymized clips for data analysis. The digital sound wave files will be achieved in the secured server at UNMC until completion of the data analysis, and then removed from the server.

Aim1: Investigators will record the swallowing sound vibrations at the anterior and posterior neck in healthy subjects, and analyze the duration, amplitude, mean frequency and power spectrum of swallowing sounds generated by various viscous foods and liquids through the pharynx.

Aim2: Investigators will compare the differences in sound duration, mean frequency and power spectrum of swallowing sounds between throat clearing and coughing in healthy subjects.

*** *** *** *** ***

Foods and Liquids Prepared for Healthy Subjects:

Foods and liquids respectively are divided into 5 levels in the International Dysphagia Diet Standardization Initiative (IDDSI) and level 3, 4 are two overlapping levels in foods and drinks Level 0 (Thin liquid) All liquid can flow through syringe Level 1 (Slightly thick liquid) There is between 1 and 4 ml remaining Level 2 (Mildly thick liquid) There is between 4 and 8 ml remaining Level 3 (Moderately thick liquid/ Liquidize) There is more than 8 ml remaining, but some liquid still flows through Level 4 (Extremely thick liquid/ Pureed) If no liquid flows at all Level 5 (Minced & Moist) Pressed with a fork the particles should easily be separated between and come through the prongs of a fork Level 6 (Soft) Sample squashes and does not return to its original shape when pressure is released.

Level 7 (Regular) No texture restrictions

Liquid Samples Preparation:

According to drink details provided in the IDDSI, investigators will choose a food polysaccharide thickener xanthan gum (UPC784672647311, Anthony's, Gluten-Free, USA) to prepare different viscous solutions. Firstly, dispersing xanthan gum in de-ionized water at 185 F for 10 min then carrying out solution in a 1.5 liter plastic beaker at 2000 rpm with a four-blade propeller (60 mm in diameter) using a 6-Speed blender (XJ-14402C, Mainstays, Walmart Inc., Bentonville, AR 72716) to ensure no lumping. After that, cool the solution to room temperature.

Flow testing: Before flow testing, we will use 10ml water flows completely through the syringe (A 10 ml slip tip syringe international standards (ISO 7886-1)) within 10 seconds to check whether the nozzle is clear and free from any plastic residue or manufacturing defects that vary occasionally occur. After checking, firstly, get a stopwatch and 2 of 10ml slip-tip syringes. Secondly, remove the plunge from one of the syringes (Syringe A). Thirdly, cover the nozzle of the syringe A with finger which makes a seal. Then using another syringe B to add the syringe A up to the 10 ml line with fluid.

According to gravity flowing test, we select the following drinks. Level 0 is de-ionized water Level 1 is xanthan gum: de-ionized water = 1oz: 5000ml Level 2 is xanthan gum: de-ionized water = 1oz: 4000ml Level 3 is xanthan gum: de-ionized water = 1oz: 3000ml Level 4 is xanthan gum: de-ionized water = 1oz: 1000ml

Food Samples Preparation:

Fork Testing: The slots/gaps between prongs of a standard metal fork are typically in 4 mm. Pressure applied to the food sample is quantified by assessment of the pressure needed to make the thumb nail blanch noticeably to white color.

According to food details provided in IDDSI, we will use IDDSI Flow Test (Syringe Test), Fork (The slots/gaps between the tines/prongs of a standard metal fork typically measure 4 mm) Drip Test and Fork Pressure Test selects food as follows:

Level 5 (Minced & Moist) cereal: de-ionized water = 2:1 Dispersing xanthan gum in de-ionized water at 185 F for 10 min then carrying out solution in a 1.5-liter plastic beaker at 2000 rpm with a four-blade propeller (60 mm in diameter) using a 6-Speed blender to ensure cereal is fully moist & minced and less than 1.5cm*1.5cm. After that, cool the solution to room temperature.

Level 6 (Soft) Banana Level 7 (Regular) White bread

ELIGIBILITY:
Inclusion Criteria:

1. Between 19-60 years old
2. Able to sign the informed consent after the whole study is explained to them
3. Self-reporting no history of swallowing disorders, neurological deficits and/or cancer of the mouth, neck or brain, or head or neck surgery
4. Able to sit upright with or without back support of chair
5. No other diseases affect swallowing function

Exclusion Criteria:

1. Have poor dentition and neurological conditions.
2. Have other diseases like cervical spondylosis, having pain when swallowing like tonsil inflammation, peritonsillar abscess, retropharyngeal abscess, pharyngeal tumor, epiglottis abscess and other diseases of the throat.
3. Have esophageal diseases such as esophageal cancers, esophageal foreign body feelings, esophagitis, etc. Neuromuscular disorders such as esophageal spasm.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participants are between 19-60 years old and able to sign the informed consent. According to self-reporting no history of swallowing disorders, neurological deficits and/or cancer of the mouth, neck or brain, or head or neck surgery, they will be able to sit upright with or without back support of chair. They have no poor dentition and neurological conditions. They don't have other diseases like cervical spondylosis, having pain when swallowing like tonsil inflammation, peritonsillar abscess, retropharyngeal abscess, pharyngeal tumor, epiglottis abscess and other diseases of the throat. They have no esophageal diseases such as esophageal cancers, esophageal foreign body feelings, esophagitis or neuromuscular disorders such as esophageal spasm.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-10-12 (Actual); Study Completion 2018-09-17 (Actual)

PRIMARY OUTCOMES:
Duration(s) of swallowing sounds among healthy subjects | 2 hours
  Investigators will record the swallowing sound vibrations at the anterior and posterior neck in health subjects, and analyze the duration(s) of swallowing sounds generated by various viscous foods and liquids through the pharynx.
Amplitude(W/m2) of swallowing sounds among healthy subjects | 2 hours
  Investigators will record the swallowing sound vibrations at the anterior and posterior neck in health subjects, and analyze the amplitude(W/m2) of swallowing sounds generated by various viscous foods and liquids through the pharynx.
Mean frequency(Hz) of swallowing sounds among healthy subjects | 2 hours
  Investigators will record the swallowing sound vibrations at the anterior and posterior neck in health subjects, and analyze mean frequency(Hz) of swallowing sounds generated by various viscous foods and liquids through the pharynx.
Power spectrum(W/Hz) of swallowing sounds among healthy subjects | 2 hours
  Investigators will record the swallowing sound vibrations at the anterior and posterior neck in health subjects, and analyze the power spectrum(W/Hz) of swallowing sounds generated by various viscous foods and liquids through the pharynx.

SECONDARY OUTCOMES:
Sound duration(s) of coughing sound and throat clearing among healthy subjects | 2 hours
  Investigators will distinguish the differences in sound duration(s) between throat clearing and coughing in healthy subjects.
Mean frequency(Hz) of coughing sound and throat clearing among healthy subjects | 2 hours
  Investigators will distinguish the differences in mean frequency(Hz) between throat clearing and coughing in healthy subjects.
Power spectrum(W/Hz) of coughing sound and throat clearing among healthy subjects | 2 hours
  Investigators will distinguish the differences in power spectrumin(W/Hz) between throat clearing and coughing in healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Chun K Siu, PhD, Study Chair — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
Acoustic analysis of swallowing sound data will be available for other researchers when all data are analyzed however voice print of IPD are not to be shared with other researchers.